CLINICAL TRIAL: NCT02951143
Title: Abuse Liability of Reduced Nicotine Content Cigarettes Within a Complex Tobacco Marketplace
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Collaborators: University of Kentucky (Other)
Responsible Party: Principal Investigator, Warren K. Bickel, Professor and Director, Virginia Polytechnic Institute and State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: R01DA042535 (NIH)
Record Dates: First submitted 2016-10-27; First posted 2016-11-01 (Estimated); Results first posted 2021-09-22 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-08

CONDITIONS: Substance-Related Disorders
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Single arm (Experimental): All participants will complete the same experimental events across 6 laboratory sessions.
  Interventions: Drug: SPECTRUM cigarettes
- 0.4 mg/g Concentration (Experimental): Participants in this arm will experience the 0.4 mg/g Concentration
  Interventions: Drug: SPECTRUM cigarettes between
- 1.3 mg/g Concentration (Experimental): Participants in this arm will experience the 1.3 mg/g Concentration
  Interventions: Drug: SPECTRUM cigarettes between
- 2.4 mg/g Concentration (Experimental): Participants in this arm will experience the 2.4 mg/g Concentration
  Interventions: Drug: SPECTRUM cigarettes between
- 5.2 mg/g Concentration (Experimental): Participants in this arm will experience the 5.2 mg/g Concentration
  Interventions: Drug: SPECTRUM cigarettes between
- 15.8 mg/g Concentration (Experimental): Participants in this arm will experience the 15.8 mg/g Concentration
  Interventions: Drug: SPECTRUM cigarettes between

INTERVENTIONS:
Drug: SPECTRUM cigarettes — Across six laboratory sessions, participants will consume 10 puffs of either their usual brand of cigarette (one session) or a SPECTRUM cigarette (five sessions) with a nicotine yield varying from 0.03 to 0.70 and either menthol (TPMF codes NRC 103, NRC 201, NRC 301, NRC 401, and NRC 601) or tobacco (TPMF codes NRC 102, NRC 200, NRC 300, NRC 400, and NRC 600) flavor, depending on preference. This will be followed by the collection of blood nicotine content and a cigarette purchase task.
  Arms: Single arm
Drug: SPECTRUM cigarettes between — Participants will be assigned one of the nicotine concentrations of a SPECTRUM cigarette. They will complete a cigarette purchase task and make real purchases for the next week. Participants will return and make purchases again, repeating 4 times.
  Arms: 0.4 mg/g Concentration; 1.3 mg/g Concentration; 15.8 mg/g Concentration; 2.4 mg/g Concentration; 5.2 mg/g Concentration

SUMMARY:
Tobacco regulatory policies can have unanticipated consequences; therefore, methods that would permit prospective estimates of the effects of potential tobacco regulations are necessary for the development of tobacco regulatory science. The goal of this project is to experimentally assess how smokers purchase and consume reduced-nicotine cigarettes. In experiment 1, we will investigate how purchasing/consuming reduced-nicotine cigarettes is related to nicotine content and absorption. In experiment 2, we will investigate how purchasing/consuming changes when other nicotine products are available in an experimental marketplace setting. The proposed projects can directly inform tobacco regulation by providing estimates of the real-world effects of novel policies.

DETAILED DESCRIPTION:
The specific objective in Experiment 1 is to examine the effect of nicotine content (0.4 mg/g, 1.4 mg/g, 2.5 mg/g, 5.6 mg/g, and 17.4 mg/g of tobacco) and blood nicotine absorption on laboratory behavioral economic measures of demand intensity and elasticity. Under double-blind conditions, we will examine the relationship between plasma nicotine and cigarette demand as a function of the dose of the nicotine in the cigarettes. Regular cigarette smokers will consume, on separate sessions, controlled puffs of a cigarette containing a blinded dose of nicotine then complete a cigarette purchase task, our measure of value, while plasma nicotine is measured. We hypothesize that cigarette demand will be associated with dose and level of circulating nicotine, but in a nonlinear fashion such that consumption of very low dose cigarettes will not be predicted by nicotine dose or intake alone.

To inform how various products may interact, we have developed and tested a novel method called the Experimental Tobacco Marketplace. The Experimental Tobacco Marketplace is a systematic extension of similar marketplace methods used with other consumer products (e.g., food marketplaces used in obesity and other nutrition-related research; Epstein, Dearing, Roba, & Finkelstein, 2010). In experimental marketplaces, multiple products are available and the experimenter controls the prices for each. These marketplaces can be either physical or virtual stores (similar to online retailers) and permit the examination of demand elasticity and intensity and degree of substitution or complementarity in consumer behavior under conditions that approximate naturalistic settings.

Experiment 2 will extend findings from the first experiment examining the effects of different concentrations of nicotine in cigarettes (0.4mg/g, 1.4mg/g, 2.5mg/g, 5.6mg/g, 17.4mg/g) and blood nictotine absorption on laboratory behavioral economic demand measures. Employing this innovative Experimental Tobacco Marketplace, we propose to examine reduced-nicotine cigarettes under the following conditions: 1) control conditions where lower dose nicotine cigarettes are the only available product in the Experimental Tobacco Marketplace and where the tobacco marketplace is similar to the current real-world marketplace (i.e., no lower dose nicotine cigarettes, but a variety of other tobacco products); 2) lower dose nicotine cigarettes are available with a number of other nicotine products excluding conventional cigarettes; and 3) lower dose nicotine cigarettes are available with a number of other nicotine products including conventional cigarettes.

ELIGIBILITY:
Inclusion Criteria:

* smoke at least 5 cigarettes per day
* have a breath carbon monoxide (CO) level of at least 10 ppm at intake
* no immediate plans to quit smoking.

Exclusion Criteria:

* pregnant, lactating, plans to become pregnant
* weigh more than 110lbs (experiment 1 only)
* have plans to move out of the area during the course of the experiment

To see if you are eligible, use the following confidential link: http://vtcri.info/arrcclinicaltrials

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 305 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2019-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Warren K Bickel, PhD, Principal Investigator — Virginia Polytechnic Institute and State University
Locations (1):
- Fralin Biomedical Research Institute at VTC, Roanoke, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Arm | 0.4 mg/g Concentration | 1.3 mg/g Concentration | 2.4 mg/g Concentration | 5.2 mg/g Concentration | 15.8 mg/g Concentration
Started | 97 | 41 | 47 | 39 | 37 | 44
Completed | 36 | 32 | 29 | 30 | 31 | 29
Not Completed | 61 | 9 | 18 | 9 | 6 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Single Arm | 0.4 mg/g Concentration | 1.3 mg/g Concentration | 2.4 mg/g Concentration | 5.2 mg/g Concentration | 15.8 mg/g Concentration | Total
Number analyzed (Participants) | 36 | 32 | 29 | 30 | 31 | 29 | 187
Age, Continuous [Mean (Inter-Quartile Range); unit: years] — Population: Each group (Various Concentrations and Single Arm) was analyzed separately.
  years
    Various Concentrations: number analyzed (Participants) | 0 | 32 | 29 | 30 | 31 | 29 | 151
    Various Concentrations |  | 41 [32.75 to 46.25] | 37 [28 to 49] | 46 [34 to 51] | 42 [36 to 51] | 39 [34 to 48] | 41 [33 to 50]
    Single Arm: number analyzed (Participants) | 36 | 0 | 0 | 0 | 0 | 0 | 36
    Single Arm | 38.5 [33 to 48.25] |  |  |  |  |  | 38.5 [33 to 48.25]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 | 12 | 16 | 15 | 13 | 87
  Male | 21 | 16 | 17 | 14 | 16 | 16 | 100
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 27 | 21 | 19 | 20 | 24 | 17 | 128
  Race: African American | 9 | 7 | 9 | 9 | 7 | 10 | 51
  Race: American Indian | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Race: More than one race | 0 | 3 | 1 | 1 | 0 | 2 | 7
Region of Enrollment [Number; unit: participants]
  United States | 36 | 32 | 29 | 30 | 31 | 29 | 187

OUTCOME MEASURES:

1. Primary Outcome: Estimated Cigarettes Taken at Free Price Derived From the Cigarette Purchase Task
Description: The Cigarette Purchase Task is a behavioral economic measure of abuse liability that consists of a series of hypothetical questions asking participants to indicate how many cigarettes they would purchase for their own consumption across a range of cigarette prices. Participants smoked one cigarette and then were asked to report how many cigarettes they would smoke within a 24 hour period at the following prices: $0.00 (free), $0.01, $0.05, $0.10, $0.25, $0.50, $1, $2, $5, $10, $25, $50, $100, $200. Nonlinear regression was then used to estimate the number of cigarettes participants would take when they were free using the equation by Koffarnus et al. (2015; doi:10.1037/pha0000045). The outcome is the logarithmically transformed number of cigarettes.
Time Frame: 10 minutes after cigarette administration
Population: Only those participants in the single arm completed this task.
Measure: Mean (Standard Error); unit: Cigarettes (log transformed)
Arm/Group | Single Arm | 0.4 mg/g Concentration | 1.3 mg/g Concentration | 2.4 mg/g Concentration | 5.2 mg/g Concentration | 15.8 mg/g Concentration
Number analyzed (Participants) | 36 | 0 | 0 | 0 | 0 | 0
Cigarettes (log transformed)
  Usual Brand | 1.50 (.0583) |  |  |  |  |
  15.8mg/g | 1.45 (.0555) |  |  |  |  |
  5.2mg/g | 1.47 (.0538) |  |  |  |  |
  2.4mg/g | 1.45 (.0678) |  |  |  |  |
  1.3mg/g | 1.37 (.0975) |  |  |  |  |
  0.4mg/g | 1.35 (.0727) |  |  |  |  |

2. Primary Outcome: Change in Blood Nicotine Content Over the Course of the Session
Description: For participants in the single arm only, blood will be collected throughout each session and analyzed for nicotine content. The change in blood nicotine content over the course of the session will be compared among the six sessions where different cigarettes were administered. Blood nicotine (expressed in ng/mL) at minute 0 was subtracted from blood nicotine at minutes 10, 15, 20, 30, 45, and 60 to yield a change in blood nicotine (negative values were truncated to 0) at each of the time points. Using these change in blood nicotine values, we calculated Area Under the Curve (AUC) via the trapezoidal rule, which resulted in a singular number (total change in blood nicotine over the course of each experimental session) in our primary outcome measure.
Time Frame: Each session (6 sessions total) with at least 2 days between each session.
Population: Only participants in the single arm had blood collected.
Measure: Mean (Standard Error); unit: ng/mL/session
Arm/Group | Single Arm | 0.4 mg/g Concentration | 1.3 mg/g Concentration | 2.4 mg/g Concentration | 5.2 mg/g Concentration | 15.8 mg/g Concentration
Number analyzed (Participants) | 36 | 0 | 0 | 0 | 0 | 0
ng/mL/session
  Usual Brand | 551.31 (24.6) |  |  |  |  |
  15.8mg/g | 350.62 (24.6) |  |  |  |  |
  5.2mg/g | 192.91 (24.6) |  |  |  |  |
  2.4mg/g | 57.11 (24.6) |  |  |  |  |
  1.3mg/g | 30.18 (24.6) |  |  |  |  |
  0.4mg/g | 6.24 (24.6) |  |  |  |  |

3. Primary Outcome: Experimental Marketplace Purchases
Description: In all arms except the single arm, measures of quantities of experimental cigarettes and other nicotine products will be obtained.
Time Frame: Sessions 2-5 with each session conducted one week apart (for 4 weeks total)
Population: This single arm did not complete the Experimental Marketplace Purchases
Measure: Mean (Standard Error); unit: grams of nicotine from non-cigarettes
Arm/Group | Single Arm | 0.4 mg/g Concentration | 1.3 mg/g Concentration | 2.4 mg/g Concentration | 5.2 mg/g Concentration | 15.8 mg/g Concentration
Number analyzed (Participants) | 0 | 32 | 29 | 30 | 31 | 29
grams of nicotine from non-cigarettes
  Current Marketplace |  | 4.07 (3.13) | 12.29 (3.47) | 15.25 (3.26) | 13.67 (3.19) | 15.25 (3.31)
  Proposed Marketplace |  | 12.70 (3.13) | 25.54 (3.47) | 17.42 (3.26) | 16.92 (3.19) | 14.93 (3.31)
  Combined Marketplace (Usual Brand Increasing) |  | 4.58 (3.13) | 11.27 (3.47) | 8.34 (3.26) | 13.30 (3.19) | 7.17 (3.31)
  Combined Marketplace (Experimental Cigarette Increasing) |  | 3.50 (3.13) | 9.62 (3.47) | 8.81 (3.26) | 11.36 (3.19) | 6.67 (3.31)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the approximately 5 weeks of participation for participants in the various concentration groups (all arms other than the single arm). Adverse event data were collected during the approximately 2 months of participation for individuals in the single arm.
Arm/Group | Single Arm | 0.4 mg/g Concentration | 1.3 mg/g Concentration | 2.4 mg/g Concentration | 5.2 mg/g Concentration | 15.8 mg/g Concentration
All-Cause Mortality (participants affected / at risk) | 0/97 | 0/41 | 0/47 | 0/39 | 0/37 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/97 | 0/41 | 4/47 | 0/39 | 2/37 | 0/44
Other Adverse Events (participants affected / at risk) | 0/97 | 0/41 | 3/47 | 0/39 | 0/37 | 1/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm (N=97) | 0.4 mg/g Concentration (N=41) | 1.3 mg/g Concentration (N=47) | 2.4 mg/g Concentration (N=39) | 5.2 mg/g Concentration (N=37) | 15.8 mg/g Concentration (N=44)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Life Events (Social circumstances) | 0 | 0 | 1 | 0 | 1 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Gall Bladder removal (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm (N=97) | 0.4 mg/g Concentration (N=41) | 1.3 mg/g Concentration (N=47) | 2.4 mg/g Concentration (N=39) | 5.2 mg/g Concentration (N=37) | 15.8 mg/g Concentration (N=44)
Life events (Social circumstances) | 0 | 0 | 0 | 0 | 0 | 1
Nausea (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Vomit after cigarette and alcohol consumption (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-11-04): https://cdn.clinicaltrials.gov/large-docs/43/NCT02951143/Prot_SAP_ICF_000.pdf